CLINICAL TRIAL: NCT02288611
Title: A Randomised, Controlled Intervention Trial to Assess the Impact of Palm Date Intake on Markers of Large Intestinal Health
Brief Title: The Impact of Palm Date Intake on Colon Health Biomarkers
Acronym: AJWA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Biochemistry, University of Reading
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AJWA STUDY
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — maltodextrin; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin/Dextrose mix (Placebo Comparator): Twenty-two healthy human individuals were randomly assigned to consume a control (maltodextrin-dextrose, 40.2g) at one of the arms period. Each arm was 21 days in duration, separated by a 14 days washout period.
  P.S. placebo is called control in this study, where the bioactive comparator is a fruit.
  Interventions: Dietary Supplement: Date fruit - Ajwa variety
- Date fruit - Ajwa variety (Active Comparator): Twenty-two healthy human individuals were randomly assigned to consume date fruits (approx. 50g) at one of the arms period. Each arm was 21 days in duration, separated by a 14 days washout period.
  Interventions: Dietary Supplement: Maltodextrin/Dextrose

INTERVENTIONS:
Dietary Supplement: Date fruit - Ajwa variety — Twenty-two healthy human individuals were randomly assigned to consume 7 date fruits (approx. 50g). Each arm was 21 days in duration, separated by a 14 days washout period.
  Other Names: Bateel Shop , London
  Arms: Maltodextrin/Dextrose mix
Dietary Supplement: Maltodextrin/Dextrose — Twenty-two healthy human individuals were randomly assigned to consume Maltodextrin/dextrose , 40.2g. Each arm was 21 days in duration, separated by a 14 days washout period.
  Arms: Date fruit - Ajwa variety

SUMMARY:
This aim of this study is to investigate the prebiotic potential of date fruits in healthy human volunteers compared to a control diet. Each arm was 21 days in duration, separated by a 14 days washout period. Faecal samples, and blood samples will be collected from each volunteer and high resolution analytical techniques (HPLC, LC-MS and NMR) will be employed to characterise the whole system metabolic response to ingestion of date fruits compared to the control. Changes in microbial parameters and metabolite profiles will be correlated with changes in biomarkers of chronic disease, including faecal water genotoxicity, cellular reactions, blood lipids and bowel movements.

DETAILED DESCRIPTION:
This aim of this study is to investigate the prebiotic potential of date fruit consumption in healthy human volunteers compared to a diet which does not contain dates; control (maltodextrin-dextrose, 40.2g) or intervention treatment 7 date fruits (50g) to 22 healthy human volunteers. Each arm was 21 days in duration, separated by a 14 days washout period. Thus, we will also address fundamental questions about the relationship between fermentation of non digestible carbohydrates, the gut microbiota and the changes in faecal short chain fatty acids (SCFA profiles), ammonia and bile acids. To this end faecal samples, and blood samples will be collected from each volunteer and high resolution analytical techniques (High Performance Liquid Chromatography; Liquid Chromatography-Mass Spectrometry and Nuclear Magnetic Resonance) will be employed to characterise the whole system metabolic response to ingestion of date fruits compared to the control. Changes in microbial parameters and metabolite profiles will be correlated with changes in biomarkers of chronic disease, including faecal water genotoxicity, cellular reactions, blood lipids and bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Body mass index - 18.5 - 30 inclusive
* Age 18 - 55 years
* Good general health as determined by medical questionnaires Requirements for diet and medication during study
* No intake of additional supplementary prebiotics (i.e. such as fructo-oligosaccharides) - please note that consumption of foods that are naturally prebiotic, e.g. cereal grains and leeks, may be consumed as normal
* No intake of probiotics (i.e. live yoghurts), drugs active on gastrointestinal motility, antibiotic treatment or any class of laxative
* All concomitant medication must be recorded in diaries and case record forms
* Usual diet, fluid intake and exercise levels should be maintained during trial period
* Please inform the investigator if you consume antibiotics during the trial. You will not be able to continue, as this may affect your faecal bacteria.

Exclusion Criteria:

* Requirements to take long-term medication active on the gastro-intestinal tract
* Use of antibiotics within the previous 6 months
* Anaemia
* Diabetes mellitus
* History of alcohol or drug abuse
* Current smoker
* Intake of any experimental drug within 4 weeks of the start of the study
* Excessive alcohol consumption (more than 21 units/wk male, 14 units/wk female)
* Females who are breast-feeding, may be pregnant, or if of child-bearing potential and are not using effective contraceptive precautions
* Major surgery, which might limit participation in, or completion of, the study.
* Participation in a study involving prebiotics or probiotics within the previous 3 months
* Physical or mental diseases that are likely to limit participation or completion of the study
* Severe allergy to foods or severe abnormal drug reactions
* Chronic gastroenterological complaints
* Intake of other supplementary prebiotics or probiotics, drugs active on gastrointestinal motility, or a laxative of any class during or within the four weeks prior to the start of the study
* Aged below 18 or over 55 years
* Have a BMI of less than 18.5 or more than 30
* Gluten allergy
* Calorie restriction or other special diet (e.g. Atkins diet, montignac diet) 6 weeks prior to the start of the study
* Vaccination against with the current season's influenza and AH1N1 flu
* Manifestation of allergy, asthma and dermatitis

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in large intestinal microbiota composition verses control intervention (0-3 months) | 3 months
  Microbial profile assessed by FISH

SECONDARY OUTCOMES:
Change from baseline in Bowel function verses the control intervention (0-3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: JEREMY PE SPENCER, PhD, Principal Investigator — UNIVERSITY OF READING - FOOD AND NUTRITIONAL SCIENCES DEPARTMENT

REFERENCES:
- [Background] Eid NM, Al-Awadi B, Vauzour D, Oruna-Concha MJ, Spencer JP. Effect of cultivar type and ripening on the polyphenol content of date palm fruit. J Agric Food Chem. 2013 Mar 13;61(10):2453-60. doi: 10.1021/jf303951e. Epub 2013 Feb 26. PMID 23406291